CLINICAL TRIAL: NCT01134718
Title: Pilot BA Study With Phase III/Commercial Versus Phase IIB Formulation. A Phase I, Open Label, Randomized, Single Dose, Crossover Study in Healthy Subjects to Assess the Relative Bioavailability of TMC435 Following Administration of Potential Phase III Formulations Compared to the Phase IIb Capsule
Brief Title: TMC435-TiDP16-C119 - A Study Comparing 2 New Capsule Formulations of TMC435 to an Established Capsule Formulation and Evaluating the Respective Blood Levels of TMC435 Following Single Dose Administration
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tibotec Pharmaceuticals, Ireland (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR017155
Record Dates: First submitted 2010-05-28; First posted 2010-06-02 (Estimated); Last update posted 2013-04-09 (Estimated); Status verified 2013-04

CONDITIONS: Hepatitis C Virus
Keywords: TMC435-TiDP16-C119; TMC435-C119; TMC435; Protease inhibitor; HCV; Hepatitis C; Bioavailability
MeSH Terms: conditions — Hepatitis C | interventions — Simeprevir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 001 (Experimental): TMC435 (F021) one morning dose of 150 mg
  Interventions: Drug: TMC435 (F021)
- 002 (Experimental): TMC435 (G006) one morning dose of 150 mg
  Interventions: Drug: TMC435 (G006)
- 003 (Experimental): TMC435 (G007) one morning dose of 150 mg
  Interventions: Drug: TMC435 (G007)

INTERVENTIONS:
Drug: TMC435 (G006) — one morning dose of 150 mg
  Arms: 002
Drug: TMC435 (F021) — one morning dose of 150 mg
  Arms: 001
Drug: TMC435 (G007) — one morning dose of 150 mg
  Arms: 003

SUMMARY:
The purpose of this study is to compare in healthy volunteers levels of TMC435 in the blood circulation after intake of 2 new capsule formulations with the level of TMC435 in the blood circulation after intake of the capsule formulation used in the Phase IIb studies.

DETAILED DESCRIPTION:
This is a randomized (study drug assigned by chance), open-label (all people involved know the treatment), single dose, crossover (volunteers will receive different treatments sequentially during the trial) study in healthy volunteers. The trial will evaluate the levels of TMC435 in the blood circulation after a single dose of 150 mg TMC435 administered as 3 different capsule formulations following breakfast. There will be a 7-day washout period between treatments and a 4-5 week follow-up at the end. Each volunteer will receive all three treatments. The main focus of the trial is the pharmacokinetic characteristics (how drugs are absorbed in the body, how they are distributed within the body and how they are removed from the body over time) of the different formulations. This evaluation requires multiple blood samples from Day 1 through 72 hours after dosing. Safety assessments (lab work, blood pressure, pulse and electrocardiogram) will follow a different schedule and are measured on Day -1 (day prior to taking first dose of drug), Day 1 (without lab work) and Day 4 of each treatment period, and 1 and 4-5 weeks after the last treatment. Each volunteer will receive 3 treatments, 7 days apart from each other. Each treatment consists of one single oral dose of 150 mg TMC435.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoker for at least 3 months
* Body Mass Index of 18.0 to 30.0 kg/m2
* Healthy based on a medical evaluation including medical history, physical examination, blood tests and electrocardiogram

Exclusion Criteria:

* Infection with Hepatitis A, B or C virus
* Infection with the human immunodeficiency virus (HIV)
* History of, or any current medical condition which could impact the safety of the participant in the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2010-06; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Rate and extent of absorption of TMC435 following administration of 3 different capsule formulations under fed condition | Measured over a period of 4 consecutive days (Day1-Day4) per treatment. Treatments (3) are 7 days apart from each other. During 1st day of each treatment, 10 blood samples for determination of pharmacokinetic characteristics are taken.

SECONDARY OUTCOMES:
All reported Adverse Events + percentage of subjects who experienced at least 1 occurrence of a given event as a measure of Safety and Tolerability following administration of single doses of 150 mg TMC435 | Till last follow up safety visit 4-5 weeks after last intake of study medication

CONTACTS AND LOCATIONS:
Overall Officials: Tibotec Pharmaceuticals Clinical Trial, Study Director — Tibotec Pharmaceutical Limited